CLINICAL TRIAL: NCT01341938
Title: Nicotine Lozenges and Assisted Self-help for Smokeless Tobacco Cessation
Acronym: LASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01CA142952 (NIH); R01CA142952-01 (NIH)
Record Dates: First submitted 2011-04-25; First posted 2011-04-26 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Smokeless Tobacco Cessation
Keywords: Smokeless Tobacco Use
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lozenge Self Help: self help materials & lozenge NRT. (Active Comparator): Self-help materials + Commit® nicotine lozenges (4 mg)
  Interventions: Drug: Commit® nicotine lozenges (4 mg) & self-help materials; Behavioral: Phone counseling & self-help materials
- Lozenge Assisted Self-help: lozenge NRT, phone counseling, & self help materials (Experimental): Self-help materials + Commit® nicotine lozenges (4 mg) + Phone counseling
  Interventions: Drug: Commit® nicotine lozenges (4 mg) & self-help materials; Behavioral: Commit® nicotine lozenges (4 mg) & phone counseling & self-help materials; Behavioral: Phone counseling & self-help materials
- Assisted Self-Help: self-help materials & phone counseling without lozenges (Experimental): Self-help materials + Phone counseling
  Interventions: Behavioral: Commit® nicotine lozenges (4 mg) & phone counseling & self-help materials; Behavioral: Phone counseling & self-help materials

INTERVENTIONS:
Drug: Commit® nicotine lozenges (4 mg) & self-help materials — Participants provided with instructions on standard use of lozenge for nicotine replacement therapy (NRT) & instructed to use the lozenge any time they have a craving or urge to use ST or tobacco. Dosing: weeks 1-6 one lozenge every 1-2 hours/16 per day, weeks 7-9 one lozenge every 2-4 hours/8 per day, weeks 10-12 one lozenge every 4-8 hours/4 per day + The "Enough Snuff" video and printed guide providing strategies for tobacco cessation.
  Other Names: Active Comparator; Lonzenge + self-help only
  Arms: Lozenge Assisted Self-help: lozenge NRT, phone counseling, & self help materials; Lozenge Self Help: self help materials & lozenge NRT.
Behavioral: Commit® nicotine lozenges (4 mg) & phone counseling & self-help materials — Three phone counseling sessions to assist in cessation from use of all tobacco + lozenge nicotine replacement therapy (NRT) + The "Enough Snuff" video and printed guide providing strategies for tobacco cessation.
  Other Names: lonzenge + phone + self-help
  Arms: Assisted Self-Help: self-help materials & phone counseling without lozenges; Lozenge Assisted Self-help: lozenge NRT, phone counseling, & self help materials
Behavioral: Phone counseling & self-help materials — Three phone counseling sessions to assist in cessation from use of all tobacco + The "Enough Snuff" video and printed guide providing strategies for tobacco cessation.
  Other Names: phone + self-help only

SUMMARY:
This research study will determine if using a combination of 4-mg nicotine lozenges, self-help materials, and/or telephone tobacco cessation counseling will help smokeless tobacco users stop using tobacco. The study will consist of three interventions:

1. The Lozenge Assisted Self-help intervention - lozenge nicotine replacement therapy, phone counseling, and self help materials
2. Assisted Self-Help intervention - self-help materials and phone counseling without lozenges
3. Lozenge Self Help intervention - self help materials and lozenge nicotine replacement therapy.

Hypothesis: The Lozenge Assisted Self-help intervention will significantly increase both the prolonged and point prevalence for all tobacco and smokeless tobacco (ST) abstinence rates at 6 months among ST users who are interested in achieving tobacco abstinence, compared to those in the Assisted Self-Help intervention and the Lozenge Self Help intervention.

DETAILED DESCRIPTION:
The overarching aim of this line of research is to develop effective ST interventions that can be disseminated. In order to accomplish our aims, the investigators will enroll 1011 ST users in a multicenter, randomized controlled trial.

The primary aims and hypotheses to be tested in this study are the following:

1. To evaluate the effectiveness of a ST intervention combining the nicotine lozenge and assisted self-help (LASH) for increasing both prolonged and point prevalence all tobacco and ST abstinence rates at 6 months follow-up compared to an assisted self-help intervention (ASH)among ST users who are interested in achieving tobacco abstinence.

   Hypothesis: The LASH intervention - adding the lozenge as nicotine replacement therapy(NRT)- will significantly increase both the prolonged and point prevalence all tobacco and ST abstinence rates compared to the ASH intervention at 6 months among ST users who are interested in achieving tobacco abstinence.
2. To evaluate the effectiveness of a ST intervention combining the nicotine lozenge and assisted self-help (LASH) for increasing both prolonged and point prevalence all tobacco and ST abstinence rates at 6 months follow-up compared to a lozenge plus self-help intervention (LSH group: no telephone counseling) among ST users who are interested in achieving tobacco abstinence.

Hypothesis: The LASH intervention will significantly increase the point prevalence abstinence rates of all tobacco and ST at 6 months compared to the LSH intervention among ST users who are interested in achieving tobacco abstinence.

Secondary aims to be tested in this study:

1. To evaluate the incremental cost-per-quit of adding the nicotine lozenge to an assisted self-help intervention (or of adding an assisted self-help intervention to a nicotine lozenge intervention)for increasing tobacco abstinence rates.
2. To evaluate changes in self-efficacy and other theoretically-relevant measures related to the use of the nicotine lozenge as potential mediators of tobacco abstinence.

The investigators will also examine an exploratory aim:

1. The primary outcome for the exploratory aim is to compare the rate of nicotine metabolism with ST abstinence. Prior research with cigarette smokers shows that the Nicotine Metabolite Ratio (NMR) [i.e., ratio of trans-3'-hydroxycotinine to cotinine) is a predictor of smoking cessation success in particular that "faster metabolizers" treated with NRT or placebo had lower quit rates compared to "slower metabolizers". The exploratory aim will test this association with Smokeless Tobacco users. The number of lozenges used is a data point to help inform this evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or over
* Currently using smokeless tobacco products as primary tobacco product
* Use smokeless tobacco for the last 6 months
* Currently want to quit
* Able to read and write English; and
* Willing to share phone number, e-mail, and mailing address with the research project
* complete informed consent process

Exclusion Criteria:

* have used behavioral or pharmacologic tobacco treatment in last 30 days
* medical history of unstable angina, myocardial infarction within the past 6 months, cardiac dysrhythmia other than medication-controlled atrial fibrillation or PSVT or medically treated or untreated hypertension with BP ≥ 180 systolic OR ≥ 100 diastolic
* have phenylketonuria (PKU)
* have another member of their household already participating in this study
* currently pregnant or nursing
* score of ≥ 15 on the Patient Health Questionnaire (PHQ-8)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1067 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Prolonged All Tobacco Abstinence | 6 months
  The primary outcome measure will be self-reported prolonged abstinence from all tobacco use at 3- and 6-month follow-up.

SECONDARY OUTCOMES:
Saliva Test for Bio-chemical Verification of Tobacco Abstinence | 6 months
  To verify self-report of prolonged abstinence, saliva will be collected once at 6 months. A salivary cotinine of < 15 ng/mL will be adjudicated as prolonged tobacco abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert H Severson, PhD, Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Insititute, Eugene, Oregon, United States

REFERENCES:
- [Result] Ebbert JO, Severson HH, Danaher BG, Benowitz NL, Schroeder DR. Nicotine Metabolite Ratio Is Associated With Lozenge Use But Not Quitting in Smokeless Tobacco Users. Nicotine Tob Res. 2016 Mar;18(3):366-70. doi: 10.1093/ntr/ntv102. Epub 2015 May 14. PMID 25977408
- [Result] Severson HH, Danaher BG, Ebbert JO, van Meter N, Lichtenstein E, Widdop C, Crowley R, Akers L, Seeley JR. Randomized trial of nicotine lozenges and phone counseling for smokeless tobacco cessation. Nicotine Tob Res. 2015 Mar;17(3):309-15. doi: 10.1093/ntr/ntu145. Epub 2014 Aug 28. PMID 25168034